CLINICAL TRIAL: NCT04698109
Title: Costituzione Della Biobanca Del Microbiota Intestinale e Salivare Umano: Dalla Disbiosi Alla Simbiosi
Brief Title: Establishment of the Human Intestinal and Salivary Microbiota Biobank - Gynecological Diseases
Acronym: BIOMIS-DIMO
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Institute of Biomembranes, Bioenergetics and Molecular Biotechnologies (Other); Istituti Tumori Giovanni Paolo II (Network); University of Bari Aldo Moro (Other); University of Salento (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMIS-DIMO
Record Dates: First submitted 2020-12-17; First posted 2021-01-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-01

CONDITIONS: Cervicovaginitis; Endometriosis; Repeated Implantation Failure
Keywords: Microbioma biobank; Biological human samples; genital system disease; Meta-omics approaches; Microbiota-pathology relationship
MeSH Terms: conditions — Endometriosis | interventions — Surveys and Questionnaires; Independent Medical Evaluation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — faeces, saliva, vaginal swab, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- recurrent cervicovaginitis: patients with recurrent cervicovaginitis
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- endometriosis: patients with endometriosis
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- repeated implantation failures: patients with repeated implantation failures
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- healthy volunteers: healthy volunteers
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination

INTERVENTIONS:
Other: Biological sample collection — Collection of faeces, urine, saliva, vaginal swab for biobanking, to evaluate the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile, and to perform routine screening
Other: Questionnaire — Anamnestic questionnaire, 3-day food questionnaire, Food Frequency Questionnaire
Other: Medical examination — Blood pressure measurement, abdominal and thoracic physical examination

SUMMARY:
This is a prospective, clinical, monocentric study aimed to collect biological samples and study microbiota from subjects suffering from subjects with recurrent cervicovaginitis, subjects with endometriosis, subjects with repeated implantation failures and from healthy volunteers. Microbiota is a complex consortium of microorganisms, located at the mucosal level (in particular intestinal, oral and vaginal) having a key role in human health and in the onset of several diseases. Microbiota alterations have been found in several diseases (gastrointestinal, metabolic, renal, oncological, gynaecological).

The study will allow to:

* Provide biological samples (faeces, saliva, vaginal, urine) from healthy volunteers and patients suffering from selected disease to the first Italian microbiota biobank;
* Study microorganisms using different in vitro and in vivo techniques;
* Study the link between the microbiota and the disease. This study is part of the BIOMIS project (Project Code: ARS01_01220), presented as part of the "Avviso per la presentazione di progetti di ricerca industriale e sviluppo sperimentale nelle 12 aree di specializzazione individuate dal PNR 2015-2020" and admitted to funding under the National Operational Program "Ricerca e Innovazione" 2014-2020 by directorial decree of MIUR - Department for Higher Education and Research - n. 2298 of 12 September 2018. BIOMIS includes several clinical studies that enrol patients with different pathologies to collect and store biological samples and study microbiota.

DETAILED DESCRIPTION:
The primary aim of this monocentric study is to populate the first national microbioma biobank with biological samples (fecal, salivary, urinary and vaginsl samples) subjects suffering from selected disease disease and healthy volunteers.

The secondary aim is the characterization of microorganisms of the biobank and study of the microbiota-pathology relationship using meta-omics, in vitro and in vivo approaches, The study plans to enrol 100 subjects at Policlinic of Bari, according to the inclusion/exclusion criteria. The study participation is voluntary, and the subjects have the right to withdraw from the study at any time and for any reason.

During the study, 3 visits are planned:

* Visit 0 (V0), including description of the objectives and procedures study, signature written informed consent, inclusion/exclusion criteria evaluation, medical examination (blood pressure measurement, abdominal and thoracic physical examination), filling in of the anamnestic questionnaire, delivery of kits for the collection of fecal, salivary and urinary material to be reported at Visit 1 and delivery of a 3-day food diary, to be completed autonomously in the days preceding the Visit 1.
* Visit 1 (V1) - at least 4 days after V0, including delivery of the of the collected biological material (feces, saliva, urine), and of a 3-day food diary, filling in of the new signs and symptoms anamnestic questionnaire and collection of the vaginal swab by medical staff.
* Telephone evaluation: administration of a "Food Frequency Questionnaire" to assess the subjects' alimentary habits.

Standard Operative Procedures (SOP) for samples storing, transport and processing will be adopted to ensure samples stability and grant results validity and quality.

Following collections, samples will be processed in different aliquots that will be used for:

* routine screening;
* storage in the first Italian human microbiote biobank (I.R.C.C.S. - Istituto Tumori "Giovanni Paolo II", Bari);
* evaluation of the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile.

Furthermore, molecular characterization of pathogenic microorganisms and pathogenic biotypes (pathovars) of commensal species of subjects with selected pathologies will be conducted.

Part of the biological material will be used for animal studies on the physiopathological role of the human intestinal microbiota transplanted into mouse models of pathology and Germ-free mouse models (specific animal study protocol developed).

The study foresees no more than minimal risk associated with blood sampling procedures. All the necessary measures to avoid any risks / inconveniences resulting from participation of the subject under study will be taken.

The study is compliant with Good Clinical Practice. Study protocol and all related documents have been approved by approved by the Independent Ethics Committees (IEC) of the involved clinical sites.

To ensure the protection and confidentiality of the participants' data, all study activities will be carried out in accordance with the European General Data Protection Regulation, Regulation (EU) 2016/679, which repeals Directive 95/46/EC.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEERS

* healthy subjects aged between 18 and 45 years, in reproductive age
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

PATIENTS WITH RECIDIVING CERVIC VAGINITIS

* healthy subjects aged between 18 and 45 years, in reproductive age
* Patients suffering from at least 3 episodes of relapsing cervicovaginitis per year: diagnosis of anaerobic vaginitis (AV) or bacterial vaginosis (BV) or vulvo-vaginal candidiasis (VVC) based on clinical symptoms and positive microscopic examination and / or positive vaginal culture
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

PATIENTS WITH ENDOMETRIOSIS

Inclusion criteria:

* aged between 18 and 45 years, in reproductive age
* patients with endometriosis: diagnosis of endometriosis carried out with transvaginal ultrasound with associated elevation of CA125
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

PATIENTS WITH REPEATED IMPLANT FAILURES (RIF)

Inclusion criteria:

* age between 18 and 45 years in reproductive age
* patients with RIF: patients who have followed PMA protocols with at least 3 failed attempts after transfer of good quality embryos
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

Exclusion Criteria:

HEALTHY VOLUNTEERS

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* HPV positive
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent onset of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* Hypertension
* eGFR (estimated glomerular filtration rate) lower than 60ml / minute and / or diagnosis of nephropathy
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Hormonal and / or intrauterine contraceptive therapy
* Healthcare workers
* Operators work with animals
* Psychiatric conditions that reduce protocol compliance.

Exclusion criteria:

POPULATION 2 - PATIENTS WITH RECIDIVING CERVIC VAGINITIS/ POPULATION 3 - PATIENTS WITH ENDOMETRIOSIS/ POPULATION 4 - PATIENTS WITH REPEATED IMPLANT FAILURES (RIF)

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent onset of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* Hypertension
* eGFR (estimated glomerular filtration rate) lower than 60ml / minute and / or diagnosis of nephropathy
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Hormonal and / or intrauterine contraceptive therapy
* Healthcare workers
* Operators work with animals
* Psychiatric conditions that reduce protocol compliance.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients with a diagnosis of recurrent cervicovaginitis, of endometriosis and subjects with repeated implantation failures attending to the clinical centres involved in the study.
  Healthy volunteers will be recruited by invitation. Enrolled subjects must not have any family relationship and hierarchical subordination with the hospitals in which biological samples will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Biological samples collection for establishment of the first National Microbiome Biobank | through study completion, an average of 1 year
  Recruitment of 100 subjects (patients with recurrent cervicovaginitis, endometriosis, repeated implantation failures and healthy volunteers) to collect biological samples for establishment of the first National Microbiome Biobank

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Cicinelli, Principal Investigator — Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari
Locations (1):
- Dipartimento di Scienze biomediche e oncologia umana (DIMO), Sezione di Ginecologia ed Ostetricia II Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma D, Chen Y, Chen T. Vaginal microbiota transplantation for the treatment of bacterial vaginosis: a conceptual analysis. FEMS Microbiol Lett. 2019 Feb 1;366(4):fnz025. doi: 10.1093/femsle/fnz025. PMID 30715301
- [Background] Yuan M, Li D, Zhang Z, Sun H, An M, Wang G. Endometriosis induces gut microbiota alterations in mice. Hum Reprod. 2018 Apr 1;33(4):607-616. doi: 10.1093/humrep/dex372. PMID 29462324
- [Background] Smith SB, Ravel J. The vaginal microbiota, host defence and reproductive physiology. J Physiol. 2017 Jan 15;595(2):451-463. doi: 10.1113/JP271694. Epub 2016 May 5. PMID 27373840
- [Background] Laschke MW, Menger MD. The gut microbiota: a puppet master in the pathogenesis of endometriosis? Am J Obstet Gynecol. 2016 Jul;215(1):68.e1-4. doi: 10.1016/j.ajog.2016.02.036. Epub 2016 Feb 18. PMID 26901277